CLINICAL TRIAL: NCT05641012
Title: Association Between Helioderma and Response to Immunotherapy in Patients With Metastatic Melanoma
Acronym: Helioma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut Jean-Godinot (Other)
Collaborators: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_HELIOMA
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Metastatic Melanoma
Keywords: metastatic melanoma; immunotherapy; helioderma; response
MeSH Terms: conditions — Melanoma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- metastatic melanoma group: adult with metastatic melanoma treated by immunotherapy
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — helioderma evaluation

SUMMARY:
Melanoma is one of the most aggressive forms of skin cancer, representing only 5% of all skin cancer but 80% of all death by skin cancer. Diagnosis and treatment of melanoma must be early because prognosis depends on stage disease.

Immunotherapy is used in metastatic melanoma. However, all patients not respond to immunotherapy.

Helioderma (photoaging) is a marker of exposure to UV rays and therefore of mutagenesis. Thus, helioderma could be associated with the response to immunotherapy.

DETAILED DESCRIPTION:
The detection and management of melanomas must be very early because the prognosis largely depends on the extent of the disease at the time of diagnosis.

For patients with melanoma, immunotherapy or dual therapy is used as treatment in unresectable and metastatic (AJCC stage IV) cases, depending on mutation status. Primary immunotherapy is possible in mutated patients in the absence of threatening progression.

However, not all patients respond well to immunotherapy, so biomarkers that predict treatment response are needed to optimize patient benefit.

The onset, development, and course of melanoma are based on the accumulation of genomic changes, including high loads of ultraviolet-induced mutations, which make melanoma the most immunogenic tumor. In several tumor types, tumor mutation load (TMB) and immune infiltration have been reported to predict response to immunotherapy. Indeed, the higher the TMB, the more the tumor is likely to produce a neo-tumor antigen, target of the reactivation of the immune system.

No threshold value of TMB has been determined to date, having a predictive value in melanoma. The degree of helioderma could be a potentially discriminating marker of the degree of UV exposure and therefore of mutagenesis. Preliminary results have reported the interest of this approach but must be confirmed because it was a small study (Russo et al).

UV-induced DNA damage results in clinical signs of heliodermia or photoaging: more or less deep wrinkles, loss of elasticity, thinning of the skin, lentigo pigmentary disorders, yellowish color of the skin, telangiectasias, on the skin areas exhibited. Helioderma could therefore be an easily accessible clinical predictor of a good response to immunotherapy.

The aim of the study is to study association between helioderma and response to immunotherapy in patients with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* metastatic melanoma
* Whatever the mutation BRAF status
* treated by immunotherapy or specific therapy
* aged more than 18
* agreeing to participate to the study

Exclusion Criteria:

* Patient whose treatment by immunotherapy has already started
* Patient who have had a radiotherapy or chemotherapy treatment
* Patient with an unknown primary melanoma, choroidal melanoma
* Patient with other cancer (except basal cell and squamous cell skin cancer)
* Patient with genetic predisposition for melanoma
* aged less than 18
* Adult not agreeing to participate to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult with metastatic melanoma treated by immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Helioderma | Day 0
  Helioderma (photoageing) evaluated around the resection scar or melanoma (if no resection) by descriptive scale ranging from 0 to 3 (3 corresponding to strong helioderma):
  * 0: no sign
  * 1: actinic lentigo, wrinkles, telangiectasia, loss of laxity, thinning
  * 2: thick, yellowish and/or dry skin, deep wrinkles, irregular pigmentation (hyper-hypopigmented spots)
  * 3: actinic keratosis, basal cell carcinoma, squamous cell carcinoma

IPD SHARING:
Plan to Share IPD: No